CLINICAL TRIAL: NCT06194162
Title: Impact of Weighted Blankets on Sleep Disturbance Among Children With Attention Deficit Hyperactivity Disorders: A Pragmatic Randomised Trial
Brief Title: Weighted Blankets for Sleep Disturbance Among Children With ADHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Collaborators: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Responsible Party: Principal Investigator, Ina Olmer Specht, Senior reseacher, University Hospital Bispebjerg and Frederiksberg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sweet Dreams
Record Dates: First submitted 2023-11-21; First posted 2024-01-08 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Attention-deficit Hyperactivity; Attention Deficit Hyperactivity Disorder; Neurodevelopmental Disorders; Sleep Disturbance; Attention Deficit Disorder; Hyperkinetic Conduct Disorder; Attention-Deficit Hyperactivity Disorder, Unspecified Type
Keywords: ADHD; weighted blanket; Children; Randomised controlled trial; Sleep Disturbance; ADD; Functional impairment
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Neurodevelopmental Disorders; Parasomnias

STUDY DESIGN:
Intervention Model Description: This study is designed as a randomised controlled trial with two parallel groups.
  Participants will be randomly assigned 1:1 into two groups using computer-generated random numbers. The allocation sequence will be stratified by age (5-8 years vs 9-12 years), ADHD medication (yes vs no) and use of melatonin/sleep medication (yes vs no).
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcome assessors will be blinded to treatment allocation where possible. Researchers will be blinded through data management and analysis. By introducing a sham blanket, participants and parents will not be made aware of their assigned intervention during the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weighted blanket (Experimental): The intervention group will receive a weighted blanket classified as a medical device class 1 as an add on to usual treatment.
  Interventions: Device: Weighted blanket
- Non-weighted blanket (Sham Comparator): The control comparator group will receive a sham intervention in the form of a non-weighted blanket. as an add on to usual treatment.
  Interventions: Device: Non-weighted blanket

INTERVENTIONS:
Device: Weighted blanket — The intervention group will receive a weighted blanket classified as a medical device class 1 as an add on to usual treatment. Participants will be asked to choose one out of at least three different weighted blankets, each with different weight classes. The choice of weighted blanket is solely taken by the participant after having tried all five blankets.
  Adherence to the weighted blanket intervention is defined as reported use 60 % of the intervention period.
  Usual treatment as part of standard care for children with ADHD, which can consist of sleep hygiene, psychoeducation, cognitive behavioral theory, medications such as melatonin or ADHD medication.
  Arms: Weighted blanket
Device: Non-weighted blanket — The control comparator will receive a sham intervention in the form of a non-weighted blanket as an add on to usual care. Participants will be asked to choose one out of two different sham blankets.
  Usual treatment as part of standard care for children with ADHD, which can consist of sleep hygiene, psychoeducation, cognitive behavioral theory, medications such as melatonin or ADHD medication.
  Arms: Non-weighted blanket

SUMMARY:
Many children with ADHD suffer from sleep disorders and dysfunction, which may affect development and well-being. According to the clinicians, some children find relief from restlessness and difficulty sleeping by using weighted blankets which have been proposed to reduce restlessness and stress via sensory integration and to calm the child by stimulating the sense of touch, muscles and joints. However, evidence for an effect on sleep is scarce, and only one RCT has investigated the effect of weighted blankets among children with ADHD. Using a RCT design, the aim is to investigate the effect on sleep disorders and dysfunction in children with ADHD aged 5-12 years by (1) using a weighted blanket during night and daytime in addition to usual treatment, compared to (2) usual treatment and a non-weighted sham blanket, with the primary outcome being differences in total sleep time. Results will support health- and social professionals who are involved in the treatment of children with ADHD.

DETAILED DESCRIPTION:
Over the past decade, interest in the relationship between sleep difficulties and ADHD has increased, with evidence showing that sleep problems are very common among school children with ADHD, affecting nearly three-quarters. Sleep problems may worsening daytime behaviors and may also affect the overall wellbeing of the family, leading to poorer parental mental health and higher stress. According to the clinicians, some children find relief from restlessness and difficulty sleeping by using weighted blankets which have been proposed to reduce restlessness and stress via sensory integration and to calm the child by stimulating the sense of touch, muscles and joints. However, evidence for an effect on sleep is scarce, and only one RCT has investigated the effect of weighted blankets among children with ADHD. Using a RCT design, the aim is to investigate the effect on sleep disorders and dysfunction in children with ADHD aged 5-12 years by (1) using a weighted blanket during night and daytime in addition to usual treatment, compared to (2) usual treatment and a non-weighted sham blanket, with the primary outcome being differences in total sleep time.

The study is designed as a superiority trial: a parallel group, randomised controlled trial, where participants are randomised to one of two study arms 1:1. The sample consists of 340 participants, divided into two groups. After randomisation each participant will stay in their assigned treatment arm during the entire study. For each study participant, the active intervention period is 28 days with assessment of primary and secondary outcomes at baseline and after 28 days of intervention. Thereafter participants will be followed through national health registers.

The trial will take place at the Child and Adolescent Mental Health Center, Mental Health Services in the Capital Region of Denmark. This center is providing assessment and treatment of children and adolescents with psychiatric disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Age 5-12 years (both included) at randomization.
3. Primary diagnosis of ADHD according to ICD-10 code F90.0, F90.1, F90.9 or F98.8.
4. Comorbidities are allowed.
5. Participated in a usual care sleep hygiene program managed by clinicians without effect within 6 months prior to enrollment.
6. If on ADHD medication or/and melatonin/sleep medication the dose must be stable, at least two weeks prior to enrollment.
7. The child and caregiver have adequate mastery of the Danish language.

Exclusion Criteria:

1. Have used any type of medical device class 1 weighted blanket before.
2. Any diagnosed diseases that markedly compromises the participant's ability to adhere to the intervention (like mental retardation, severe underweight, chronic respiratory or circulatory conditions, surgical implants, osteoporosis).
3. Another member of the household enrolled in the trial.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 340 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Changes in total sleep time (average minutes per day) | Week 0 and 4
  Total sleep time (TST) is defined as the time of total sleep episode minus the awake time (the entire time spent sleeping) and reported in minutes per day. TST per day will be measured using actigraphy in form of MotionWare 8 (The MotionWare 8®-CamNtech MotionWare).

SECONDARY OUTCOMES:
Changes in functional impairment | Week 0 and 4
  Functioning impairment will be measured using Weiss Functional Impairment Rating Scale (WFIRS-P). The WFIRS-P is a 50-item scale assessment tool where caregivers rate the impact of their child's emotional or behavioural problems in the previous month on six separate domains: (A) Family (ten items); (B) School and learning; (C) Life skills; (D) Child's self-concept; (E) Social activities; and (F) Risky activities. Each item is rated on a four-point scale from 0 ('never or not at all') to 3 ('very often or very much') or rated as 'not applicable'. The instrument uses a likert scale such that any item rating 2 or 3 is clinically impaired. The mean of all scored items for each domain will be calculated. Furthermore, a single overall WFIRS-P score will also be calculated as the average of the six domain scores.
Changes in sleep onset latency (average minutes per day) | Week 0 and 4
  Sleep onset latency (SOL) refers to the period of time between turning lights out to go to sleep and falling asleep. SOL will be measured using actigraphy which includes a button that should be pressed by a caregiver when the lights are turned off. SOL will be reported as minutes per day.
Changes in number of awakenings (numbers per night) | Week 0 and 4
  Wake after sleep is defined as number of minutes scored as wake during sleep period and will be measured using actigraphy.
Changes in sleep efficiency (percentage) | Week 0 and 4
  Sleep efficiency (SE) is measured using actigraphy and is the actual sleep time expressed as a percentage of the total time in bed (the time elapsed between "lights out" and "get up time"). SE will be reported as minutes per day.
Changes in ADHD core symptoms (score point) | Week 0 and 4
  ADHD core symptoms will be measured with Attention Deficit Hyperactivity Disorder Rating Scale (ADHD-RS) parent version. It is a 26-item questionnaire including the 18 original ADHD-RS-IV items supplied with 8 conduct problem items. All items are rated on a 4-point Likert scale (0-3), where 0 represents never or rarely, 1 is sometimes, 2 is often, and 3 is very often. From the item scores, a total score ranging 0-78 will be calculated. Further, three sub-scores will be calculated; inattentive scale: range 0-27, hyperactive/impulsive scale: range 0-27, and conduct scale: range 0-24.
Changes in parental stress (score point) | Week 0 and 4
  Changes in parental stress is measured by the Parental Stress Scale (PSS). The PSS is an 18-item questionnaire assessing parents' feelings about their parenting role, exploring both positive aspects (e.g. emotional benefits, personal development) and negative aspects of parenthood (e.g. demands on resources, feelings of stress). Parents can agree or disagree in terms of their typical relationship with their child or children. Responses are scored as follows: strongly disagree, disagree, undecided, agree, strongly agree. To compute the parental stress score, items 1, 2, 5, 6, 7, 8, 17, and 18 should be reversely scored as follows: (1=5) (2=4) (3=3) (4=2) (5=1). The item scores are then summed. Parental stress scores range from 18 to 90, with lower scores indicating lower levels of parental stress.
Changes in child quality of life (score point) | Week 0 and 4
  Child quality of life will be measured using The World Health Organisation- Child Well-Being Index (WHO-5). The WHO-5 Child Wellbeing Index is a simple self-reported measure of children's psychological wellbeing. The tool consists of five statements describing a positive state. The child is asked to say how often they felt that way during the past two weeks, by selecting one of the following options: All the time, Often, Sometimes, Rarely or Never.
Adverse events (Number of participants with adverse events) | During intervention
  Number of participants with adverse events (AE).
Serious adverse events (Number of participants with serious adverse events) | During intervention
  Number of participants with serious adverse events (SAE).

OTHER OUTCOMES:
Changes in sensory modulation disorder (score point) | Week 0 and 4
  Changes from baseline to end of treatment in the caregiver-rated Sensory Processing Measure 2 (SPM-2). The 80 likert-type items include eight different scales: social participation, vision, hearing, touch, taste and smell, body awareness, balance and motion and finally planning and ideas, which capture related but separate aspects of sensory processing difficulties. Responses never, occasionally, frequently, or always correspond to the numeric values 1 to 4 respectively, to indicate the frequency of behaviors. A total raw score is calculated with a higher score suggesting greater dysfunction. Raw scores are also converted to T-scores and percentile scores that can fall into three ranges. T-scores in the range of 40 to 59 represent Typical functioning, T-scores in the range of 60 to 69 represent moderate difficulties in functioning, and T-scores of 70 or above represent severe difficulties in functioning.
Cost effectiveness | Week 0 and 4
  Assessed by health economic aspects, such as quality-adjusted life year (QALY) and productivity loss among caregivers.
Changes in functional impairment | 2 years after end of treatment.
  Functioning impairment will be measured using Weiss Functional Impairment Rating Scale (WFIRS-P). The WFIRS-P is a 50-item scale assessment tool where caregivers rate the impact of their child's emotional or behavioural problems in the previous month on six separate domains: (A) Family (ten items); (B) School and learning; (C) Life skills; (D) Child's self-concept; (E) Social activities; and (F) Risky activities. Each item is rated on a four-point scale from 0 ('never or not at all') to 3 ('very often or very much') or rated as 'not applicable'. The instrument uses a likert scale such that any item rating 2 or 3 is clinically impaired. The mean of all scored items for each domain will be calculated. Furthermore, a single overall WFIRS-P score will also be calculated as the average of the six domain scores.
Changes in ADHD core symptoms (score point) | 2 years after end of treatment.
  ADHD core symptoms will be measured with Attention Deficit Hyperactivity Disorder Rating Scale (ADHD-RS) parent version. It is a 26-item questionnaire including the 18 original ADHD-RS-IV items supplied with 8 conduct problem items. All items are rated on a 4-point Likert scale (0-3), where 0 represents never or rarely, 1 is sometimes, 2 is often, and 3 is very often. From the item scores, a total score ranging 0-78 will be calculated. Further, three sub-scores will be calculated; inattentive scale: range 0-27, hyperactive/impulsive scale: range 0-27, and conduct scale: range 0-24.
Changes in parental stress (score point) | 2 years after end of treatment.
  Parental stress is measured by the Parental Stress Scale (PSS). The PSS is an 18-item questionnaire assessing parents' feelings about their parenting role, exploring both positive aspects (e.g. emotional benefits, personal development) and negative aspects of parenthood (e.g. demands on resources, feelings of stress). Parents can agree or disagree in terms of their typical relationship with their child or children. Responses are scored as follows: strongly disagree, disagree, undecided, agree, strongly agree. To compute the parental stress score, items 1, 2, 5, 6, 7, 8, 17, and 18 should be reversely scored as follows: (1=5) (2=4) (3=3) (4=2) (5=1). The item scores are then summed. Parental stress scores range from 18 to 90, with lower scores indicating lower levels of parental stress.
Changes in child quality of life (score point) | 2 years after end of treatment.
  Child quality of life will be measured using The World Health Organisation- Child Well-Being Index (WHO-5). The WHO-5 Child Wellbeing Index is a simple self-reported measure of children's psychological wellbeing. The tool consists of five statements describing a positive state. The child is asked to say how often they felt that way during the past two weeks, by selecting one of the following options: All the time, Often, Sometimes, Rarely or Never.
Cost effectiveness | 2 years after end of treatment.
  Assessed by health economic aspects, such as quality-adjusted life year (QALY) and productivity loss among caregivers.

CONTACTS AND LOCATIONS:
Overall Officials: Ina O. Specht, Ph.d., Principal Investigator — Research Unit for Dietary Studies, The Parker Institute
Locations (1):
- The Parker Institute, Bispebjerg and Frederiksberg Hospital, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rohde JF, Ginnerup-Nielsen E, Larsen SC, Tjott C, Christensen R, Heitmann BL, Waehrens EE, Pagsberg AK, Specht IO. Impact of weighted blankets on sleep disturbance among children with attention deficit hyperactivity disorders (ADHD): study protocol for a pragmatic randomised controlled trial. BMC Psychiatry. 2025 Apr 8;25(1):345. doi: 10.1186/s12888-025-06768-6. PMID 40200167